CLINICAL TRIAL: NCT07336290
Title: One-stop Evaluation of Hypertrophic Cardiomyopathy in Cardiac Magnetic Resonance
Status: Enrolling by invitation | Type: Observational
Sponsor: Minjie Lu (Other)
Responsible Party: Sponsor-Investigator, Minjie Lu, Principal Investigator, Chinese Academy of Medical Sciences, Fuwai Hospital
Organization: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Other Study IDs: One-stop HCM
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-01

CONDITIONS: Hypertrophic Cardiomyopathy (HCM)
Keywords: cardiac magnetic resonance; diagnosis; risk stratificaiton; artificial intelligence; personalized prognosis
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hypertrophic myocardium

SUMMARY:
This is a multi-center, observational study aiming to establish a precision diagnosis scheme and multi-dimensional risk prediction models for Hypertrophic Cardiomyopathy (HCM). The study plans to enroll 10000 adult HCM patients. It will integrate genetic testing, advanced cardiac imaging (echocardiography and cardiac magnetic resonance), and biomarker analysis to develop early diagnosis, differential diagnosis, and new risk prediction models for sudden cardiac death (SCD) and heart failure in HCM patients. Participants will undergo baseline assessments and be followed up every six months for up to 3 years to track clinical outcomes. This study is non-interventional and does not involve any investigational drugs or devices.

ELIGIBILITY:
Inclusion Criteria:

A maximal left ventricular wall thickness of ≥ 12 mm in any segment at end-diastole, as measured by echocardiography or Cardiac Magnetic Resonance (CMR)

Exclusion Criteria:

* Presence of any contraindication to CMR examination.
* Unwillingness to participate in the study or to provide informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with hypertrophic myocardium experienced CMR scanning
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2028-07-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with sudden cardiac death | 5-year

SECONDARY OUTCOMES:
Number of participants with all-cause mortality | 5-year
Number of participants with atrial fibrillation | 5-year
Number of participants with heart failure hospitalization | 5-year